CLINICAL TRIAL: NCT07350382
Title: Development and Internal Validation of a Machine Learning-Enhanced Nomogram to Stratify Risk of Chronic Cognitive Impairment Following Pediatric Posterior Fossa Surgery
Brief Title: Predicting Cognitive Dysfunction After Pediatric Posterior Fossa Tumor Surgery
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Lan, Professor, West China Hospital
Other Study IDs: WestChinaH-HX-2025-012
Record Dates: First submitted 2026-01-05; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2024-01

CONDITIONS: Posterior Fossa Tumors; Pediatric Tumor of Brain
Keywords: Pediatric posterior fossa tumor; Cognitive dysfunction; Cerebellar cognitive affective syndrome; Predictive model; Machine learning; Nomogram; Calibration curve
MeSH Terms: conditions — Infratentorial Neoplasms; Cognitive Dysfunction; Cerebellar Cognitive Affective Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric patients who underwent surgical resection of a posterior fossa tumor: Stratify this cohort into two subgroups based on outcome:
  Those with long-term cognitive dysfunction (n=172) Those without (n=428)
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study

SUMMARY:
The goal of this observational study is to develop and validate a clinical prediction model to identify risk factors for long-term cognitive dysfunction in children (ages 0-18 years) who have undergone surgical resection of a posterior fossa tumor. The main questions it aims to answer are:

Can a combination of preoperative and postoperative clinical, surgical, and neuroimaging factors accurately predict which children will develop long-term cognitive dysfunction after posterior fossa tumor surgery? Is white matter integrity-specifically fractional anisotropy (FA) of the superior cerebellar peduncle (SCP)-a key independent predictor of cognitive outcomes? Researchers will compare children who developed long-term cognitive dysfunction (cases) to those who did not (controls) to see if differences in imaging biomarkers (e.g., SCP FA, fMRI abnormalities), tumor characteristics (e.g., location, volume, histology), treatment factors (e.g., radiotherapy, surgical approach), and demographic variables (e.g., age) are associated with cognitive outcomes.

Participants were not asked to perform any tasks or receive any interventions as part of this study, because it is a retrospective analysis of existing medical records and imaging data. Data collected included:

Preoperative and postoperative brain MRI and DTI scans Tumor pathology and surgical reports Treatment details (e.g., radiation, chemotherapy) Neuropsychological assessment results at 1-year follow-up

ELIGIBILITY:
Inclusion Criteria:

* Age 0-18 years at time of surgery
* Histopathologically confirmed primary posterior fossa tumor (e.g., medulloblastoma, ependymoma, pilocytic astrocytoma)
* Underwent surgical resection of the tumor at the hospital
* Availability of preoperative brain MRI and diffusion tensor imaging (DTI)
* Completed standardized neuropsychological assessment at approximately 1 year post-surgery

Exclusion Criteria:

* Pre-existing neurological or neurodevelopmental disorders (e.g., autism, intellectual disability, cerebral palsy)
* History of prior cranial irradiation or chemotherapy before posterior fossa surgery
* Incomplete clinical, imaging, or follow-up data required for model variables
* Tumor recurrence or progression before 1-year cognitive assessment
* Non-posterior fossa primary brain tumors (e.g., supratentorial gliomas)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study includes 600 children aged 0-18 years who underwent surgical resection of a primary posterior fossa tumor (e.g., medulloblastoma, ependymoma, or pilocytic astrocytoma). All participants had preoperative brain MRI with diffusion tensor imaging (DTI), received standard-of-care treatment, and completed comprehensive neuropsychological assessments at approximately 1 year post-surgery. The cohort represents a real-world pediatric neuro-oncology population treated at multiple tertiary care centers.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Long-Term Cognitive Dysfunction | 1 year
  Presence or absence of long-term cognitive dysfunction, defined as a full-scale IQ (FSIQ) score < 85 or significant impairment in ≥2 cognitive domains (e.g., attention, memory, executive function, processing speed) on standardized neuropsychological assessment at 1-year follow-up.

SECONDARY OUTCOMES:
Model Discrimination Performance | 1 year post-surgery
  Area Value under the receiver operating characteristic curve (AUC) of the final predictive model (nomogram) in the internal validation cohort.
Model Calibration Accuracy | 1 year after surgery
  Agreement degree between predicted probability and observed frequency of cognitive dysfunction, assessed by Hosmer-Lemeshow test P Value.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol